CLINICAL TRIAL: NCT00194298
Title: FDG-PET Imaging in Complicated Diabetic Foot (Protocol Version Dated 3/01/2004)
Brief Title: FDG-PET Imaging in Complicated Diabetic Foot
Status: Active, not recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: R01DK063579-04 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Diabetic Foot Disease
Keywords: diabetic foot disease; osteomyelitis; charcot; neuropathy; hypoxia; [18 F] Fluorodeoxyglucose; Positron Emission Tomography Imaging
MeSH Terms: conditions — Osteomyelitis; Hypoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Procedure: FDG-PET Imaging

SUMMARY:
The main objective of the proposed research study is to determine the potential utilization of [18-F] Fluorodeoxyglucose (FDG) positron emission tomography (PET) in patients with complicated diabetic foot, especially in the diagnosis or exclusion of osteomyelitis in this setting. We intend to validate and establish the necessary criteria for making such a diagnosis and determine the accuracy of the technique through comparison with other existing modalities, including MRI, and patient outcome. We expect that at the completion of the proposed research, the role of these powerful imaging modalities will be clearly defined in the management of patients with this challenging and serious complication.

DETAILED DESCRIPTION:
FDG-PET imaging is a promising imaging technique, which has the potential to overcome many of the shortcomings mentioned previously with regard to radiologic and scintigraphic methodologies. FDG is a diagnostic tracer utilized to measure the metabolic rates of normal and abnormal tissues. Many investigators have noted the affinity of FDG for active inflammatory and infectious disorders, such as sarcoidosis, the abdominal abscess, brain abscess, lung abscess, renal abscess, inflammatory pancreatic disease, lobar pneumonia, asthma, tuberculosis, colitis, sinusitis, myositis, mastitis, vasculitis, deep venous thrombosis, thyroiditis and other infections including those encountered in orthopedic patients.

According to the literature, the most accurate nuclear medicine modality for detecting infection associated with diabetic foot is the labeled WBC method. We hypothesize that FDG-PET imaging has several advantages over this method. Detection of infection by labeled WBC imaging is based upon the assumption that the administered cells will migrate to the sites of infection. Since the majority of the labeled leukocyte preparation consists of neutrophils, inflammatory/infectious processes with a predominantly neutrophilic infiltrate (acute infections) are likely to yield positive results. However, most infections associated with diabetic foot are sub-acute or chronic. Consequently, the dominant inflammatory cells involved are monocytes and lymphocytes. Therefore, labeled leukocytes are unlikely to detect chronic infection since very few monocytes and lymphocytes are labeled. In addition, the previous treatment (antibiotics, etc) can severely reduce the chemotropic effect of bacteria and therefore, fewer leukocytes will migrate to the infectious sites, rendering the labeled leukocyte method ineffective.

In contrast, the uptake of FDG in inflammatory cells reflects "in vivo labeling" of the existing cells at the site of infection soon after the administration of the compound. This would indicate that FDG-PET technique might allow imaging a substantially larger population of cells, which are residing in the area of infection and inflammation. Therefore, in addition to considerable simplification of procedures associated with the labeled WBC method, including the time required to complete the study, this approach may provide higher sensitivity for diagnosing infection in such settings. Furthermore, since FDG uptake does not rely upon leukocyte migration, treatment with antibiotics is less likely to affect its sensitivity in delineating the sites of infection. One possible advantage of the labeled WBC method over FDG-PET imaging is that high serum glucose levels do not appear to have an adverse effect on the test results with the former technique while hyperglycemia is known to decrease tumor cell FDG uptake. However, our preliminary results indicate that high glucose levels do not negatively affect FDG uptake by inflammatory cells. Based on these observations, FDG-PET imaging appears to be an attractive alternative to conventional techniques for the detection of infection.

FDG-PET imaging offers a unique tool for the diagnosis and management of the diabetic foot. Through the establishment of appropriate diagnostic criteria, a PET scan may prove to be highly accurate in localizing deep infections of bone and soft tissue associated with the complicated diabetic foot. By distinguishing these infections from inflammation, it has the potential to become the optimal diagnostic imaging technique with which to diagnose and manage patients with diabetic foot. Therefore, research studies designed to further validate the ability of this technique are essential to achieving this goal.

ELIGIBILITY:
Inclusion Criteria:

* The 240 patients selected for entry into this study will be men or women of any ethnic background diagnosed with diabetic foot disease by members of the team in the Diabetes Center of the Department of Medicine and the division of Vascular Surgery of the department of Surgery at the University of Pennsylvania Health System (Hospital of the University of Pennsylvania).

Study I: FDG-PET imaging of patients with diabetic foot without clinical suspicion of osteomyelitis or deep-seated tissue infections The patients must have clinical diagnosis of uncomplicated diabetic foot. Each patient will undergo appropriate evaluation including history, physical examination, standard radiographic evaluation (including MRI), and grading of peripheral neuropathy using the Michigan Neuropathy Screening Instrument (MNSI). Patients will be divided into three groups, corresponding to MNSI score of 0-3, 4-8, and 9-13, which we will classify as mild, moderate, and severe, respectively. We intend to enroll 26 patients in each of the first two groups and 27 patients in the third.

Study II: FDG-PET imaging of patients with diabetic foot and clinical suspicion of osteomyelitis or deep-seated infections The patients must have clinical diagnosis of complicated diabetic foot. These patients will be those suspected of having a deep-seated infection and may or may not be scheduled to undergo amputation or debridement of affected tissue. Each patient will undergo an appropriate evaluation including history, physical examination, radiologic examination including MRI, MNSI, and vascular assessment by segmental Doppler pressures and pulse wave recording.

Exclusion Criteria:

* Patients with complications of the foot with etiologies not related to diabetes will be excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 240 patients selected for entry into this study will be men or women of any ethnic background diagnosed with diabetic foot disease and/or patients with diabetes and suspected infection(s) below the hip by members of the Diabetes Center of the Department of Medicine, the Division of Vascular Surgery of the Department of Surgery at the University of Pennsylvania Health System (Hospital of the University of Pennsylvania), the Ankle and Foot Medical Centers of Delaware Valley (PENN Presbyterian Hospital, and the Pennsylvania Orthopedic Foot and Ankle Surgeons (Pennsylvania Hospital).
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2002-10; Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
SUV measurement from PET scan | Following completion of PET scan
  Standardized Uptake Value

CONTACTS AND LOCATIONS:
Overall Officials: Abass Alavi, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States